CLINICAL TRIAL: NCT01525355
Title: A Prospective Study Evaluation the Role of EUS Prior to ERCP in the "Positive" Setting of Positive Intraoperative Cholangiogram (IOC) During Cholecystectomy
Brief Title: EUS Prior to ERCP in the Positive Setting of Positive Intraoperative Cholangiogram (IOC) During Cholecystectomy
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00013737
Record Dates: First submitted 2012-01-30; First posted 2012-02-02 (Estimated); Last update posted 2017-11-07 (Actual); Status verified 2017-04

CONDITIONS: Calculi; Stenosis of Bile Duct
Keywords: EUS; ERCP; Intraoperative cholangiogram; Cholecystectomy; Common Bile Duct Stones; Strictures; Stenosis; Duodenum; Dilated Bile duct; Non-filling of the duodenum by contrast
MeSH Terms: conditions — Calculi; Constriction, Pathologic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- EUS prior to ERCP

SUMMARY:
Performing an EUS prior to ERCP in the setting of a positive intraoperative cholangiogram will identify and risk stratify patients for the presence of CBD stones and strictures.

DETAILED DESCRIPTION:
During routine cholecystectomy, surgeons will often perform an intraoperative cholangiogram in an effort to define anatomical landmarks and ensure patency and drainage of the common bile duct. This involves injecting a radiopaque contrast medium into the biliary tree during the operation. Occasionally contrast injection onto the common bile duct will reveal an abnormality and are deemed a "positive intraoperative cholangiogram" (positive IOC). These abnormalities can include the following: single or multiple stones; non-filling of the duodenum by contrast; stenosis or narrowing of the common bile duct (CBD). When discovered these findings are better addressed and treated endoscopically via endoscopic retrograde cholangiopancreatography (ERCP). ERCP's are considered the gold standard for the diagnosis and treatment of positive intraoperative cholangiograms. However, several studies have shown that 40-50% of patients who undergo an ERCP after a "positive" IOC have a normal cholangiogram. Reasons for this include spontaneous stone passage of the stone, dysmotility of the biliary tree, or poor quality, incomplete, or misinterpretation of the IOC. Therefore ERCP's are being performed when they could be avoided. ERCP performance carries significant complications including pancreatitis (5-10%), bleeding, and perforation. Ideally if a safer test to assess the bile duct could be performed immediately prior to the ERCP to confirm the presence of the positive IOC findings, this would ensure that the ERCP is being performed for therapeutic means thus avoiding unnecessary ERCP's.

EUS is often performed prior to ERCP's under the same sedation in our endoscopy unit. From 2005 to 2007, two hundred and twenty seven "combined EUS and ERCP procedure were performed.(unpublished internal data). Our experience with "combined" EUS and ERCP procedures has demonstrated that performing an EUS prior to an ERCP will prolong the total procedure time less than 10 minutes with no significant increase in adverse events. Performance of an EUS prior to ERCP to confirm biliary pathology after a "positive" IOC has never been studied in a rigorous fashion.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be able to review and sign informed consent
* Cholecystectomy must have been performed within one month of enrollment
* Positive intraoperative cholangiogram
* Stone
* Multiple Stones
* Stenosis
* "non filling" of duodenum
* Dilated bile duct

Exclusion Criteria:

* Cannot give and sign informed consent

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who have gone an uncomplicated cholesytectomy and determined to have a "positive intraoperative cholangiogram" within one month of presentation to Wake Forest Baptist Health.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2010-10 (Actual); Primary Completion 2016-06-07 (Actual); Study Completion 2016-06-07 (Actual)

PRIMARY OUTCOMES:
Bile Duct | 2 years
  Stone seen by EUS confirmed by ERCP

SECONDARY OUTCOMES:
Lesions | 2 Years
  Presence of obstuctinn lesion seen by EUS
Bile duct | 2 years
  Diameter of common bile duct and common hepatic duct
Diverticulum | 2 years
  Presence of periampullary diverticulum seen by endoscopy
ERCP | 2 years
  Number of ERCP's that could have been avoided
ERCP | 2 years
  Complications from ERCP

CONTACTS AND LOCATIONS:
Overall Officials: John A Evans, MD, Principal Investigator — Wake Forest University Baptist Health
Locations (1):
- Wake Forest Baptist Health, Winston-Salem, North Carolina, United States